CLINICAL TRIAL: NCT02575326
Title: Developing Patient-Centered Approaches to Asthma Management in Obese Adolescents
Brief Title: Teen Asthma Control Encouraging a Healthier Lifestyle
Acronym: TAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Christine Joseph, Senior Epidemiologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8298
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-02

CONDITIONS: Asthma; Obesity
Keywords: Asthma, Body Mass Idex, BMI, Overweight, Obesity
MeSH Terms: conditions — Asthma; Obesity; Overweight

STUDY DESIGN:
Masking Description: Physicians are randomized. Eligible youth that present to the participating physician assume the assignment of that physician
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Control (Other): Teens in the control group will receive standard or usual care as provided by their physician.
  Interventions: Other: Standard Control
- Intervention (Other): Teens in the intervention group will receive a provider administered, tailored discussion guide based on motivational interviewing techniques.
  Interventions: Behavioral: a provider administered, tailored discussion guide

INTERVENTIONS:
Other: Standard Control — Teens in the control group will receive standard or usual care as provided by their physician.
  Arms: Standard Control
Behavioral: a provider administered, tailored discussion guide — Teens in the intervention group will receive a provider administered, tailored discussion guide based on motivational interviewing techniques.
  Arms: Intervention

SUMMARY:
Little guidance is given to physicians caring for obese adolescents with asthma, however, findings suggest that interventions designed to achieve asthma control in these patients are necessary. Because of the psychosocial factors often associated with obesity and asthma (e.g., low self-esteem, depression, and low quality of life) successful interventions should incorporate a patient-centered approach. The proposed study design is a clinic-based, randomized controlled trial (RCT) in teens with a history of asthma and who are overweight or obese.

DETAILED DESCRIPTION:
Asthma that has persisted in adolescents is likely to persist into adulthood. For 25-30% of Americans, adolescence is also the period at which they experience their greatest weight gain, particularly as they approach the final stages of puberty. Asthma management may be more of a challenge in the overweight adolescent compared to a normal weight youth. Asthma related morbidity is increased in overweight patients, reflected in higher health care utilization for this subgroup. Little guidance is given to physicians caring for obese adolescents with asthma, but findings suggest that interventions designated to achieve control in these patients are necessary. Because of the psychosocial factors often associated with obesity and asthma (e.g. low self-esteem, depression and low quality of life) successful interventions should incorporate a patient-centered approach.

Patient-centered care (or patient focused care) involves a partnership between the patient and the physician, shared discussion making, as well as productive communication and health promotion. The objective of this project is to collect the information necessary to develop a tailored discussion guide for use by the physician caring for the obese teen with asthma. Project results will provide an evidence base for the development and evaluation of additional patient-centered health interventions for obese adolescents with asthma. The investigators will conduct this study among patients whom eligibility can be determined using the electronic medical record (EMR). The specific aims of this proposal are to:

Qualitatively collect information on outcomes important to obese adolescents with asthma:

Create a tailored discussion guide that incorporates patient preferences and treatment goals that can be used by providers caring for overweight adolescents with asthma:

Conduct a randomized trial to determine if patient-centered and clinical outcomes improve for patients whose physicians use the tailored discussion guide compared to those who do not.

ELIGIBILITY:
Inclusion Criteria:

* BMI >85th Percentile & Diagnosed with asthma; using a modification of Healthcare Effectiveness Data and Information Set (HEDIS) criteria:
* At least one emergency department visit with a principal diagnosis of asthma, or
* At least one acute inpatient claim/encounter with asthma as the principal diagnosis or at least four outpatient visits with an asthma diagnosis and at least or
* At least four asthma four outpatient visit with an asthma diagnosis and at least two asthma medications dispensed, or
* At least four asthma medications dispensed in the last 12 month

Exclusion Criteria:

* Does not meet eligibility criteria for weight and/or asthma;
* Currently enrolled in another investigational asthma management /education/weight management trial.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2015-08; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test | 12 months of enrollment
  A validated measure of asthma control

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 12 months of enrollment
  changes in participant weight

CONTACTS AND LOCATIONS:
Overall Officials: Christine Joseph, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Joseph CLM, Alexander GL, Lu M, Leatherwood SL, Kado R, Olden H, Melkonian C, Miree CA, Johnson CC. Pilot study of a brief provider and EMR-based intervention for overweight teens with asthma. Pilot Feasibility Stud. 2021 Aug 30;7(1):167. doi: 10.1186/s40814-021-00848-6. PMID 34462008